CLINICAL TRIAL: NCT04873050
Title: A Randomized, Placebo-controlled, Double Blind Trial of Semaglutide 1mg (Ozempic®) on Regression to Normoglycemia in WomEn with a Recent History of Gestational DiabETes Mellitus: the SWEET Study
Brief Title: Treatment to Regress to Normoglycemia in Women with a Recent History of GDM
Acronym: SWEET
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Woman's (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Principal Investigator, Elizabeth F Sutton, PhD, Director of Scientific Research, Woman's
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RP-21-010
Record Dates: First submitted 2021-04-29; First posted 2021-05-05 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Pre Diabetes; Postpartum Disorder
MeSH Terms: conditions — Glucose Intolerance; Puerperal Disorders | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Semaglutide Pen Injector (Ozempic) (Experimental): Weekly injections of semaglutide for 8 months total (2 months of titration; 6 months of full dose- 1mg/week)
  Interventions: Drug: Semaglutide Pen Injector [Ozempic]
- Placebo (Sham Comparator): Weekly injections of placebo for 8 months total
  Interventions: Drug: Placebo semaglutide pen injector

INTERVENTIONS:
Drug: Semaglutide Pen Injector [Ozempic] — Start injection of semaglutide 0.25mg subcutaneously (SC) once a week for 4 weeks; step up to 0.5 mg SC QD for once a week for 4 weeks to a final dose of 1.0 mg semaglutide SQ weekly for 24 doses
  Other Names: Semaglutide 1mg; Ozempic
  Arms: Semaglutide Pen Injector (Ozempic)
Drug: Placebo semaglutide pen injector — Start injection of placebo semaglutide 0.25mg subcutaneously (SC) one a week for 4 weeks; step up to 0.5 mg SC QD for once a week for 4 weeks to a final dose of 1.0 mg semaglutide SQ weekly for 24 doses
  Other Names: Placebo Semaglutide 1mg; Placebo Ozempic
  Arms: Placebo

SUMMARY:
The purpose of the study is to determine the efficacy of semaglutide 1mg (Ozempic®) to aid recently postpartum women with dysglycemia and a history of GDM to regress to normoglycemia; thereby filling a gap in efficacious pharmacologic intervention options for clinicians to support postpartum diabetes recovery and reduce future risk of T2DM in young women.

DETAILED DESCRIPTION:
The diagnosis of gestational diabetes mellitus (GDM) during pregnancy identifies young women with abnormalities in pancreatic beta cell function that worsen over time, leading to diabetes. It is estimated that between 15% and 70% of women with a history GDM will progress to type 2 diabetes mellitus (T2DM). However, upon an impaired glucose tolerance test result in the early postpartum period, the American College of Obstetricians and Gynecologists only recommend considering referral for management, weight loss and physical activity counseling, considering metformin if testing results are severe enough, and yearly assessment of glycemic status. In many cases, it is possible to reverse diabetes by losing weight in the early stages before permanent, systemic damage occurs. Therefore, there is a dire need for efficacious pharmacologic intervention options in this period of postpartum diabetes recovery to return women to normoglycemia and lower future T2DM risk. Weight loss and medications that mitigate impairments in insulin secretion show the best promise for delaying or preventing T2DM, the dominant form of diabetes that develops after GDM. The primary study objective is "to examine the efficacy of semaglutide 1mg compared to placebo on regression to normoglycemia in women with dysglycemia and a recent history of gestational diabetes mellitus (i.e., 6-36 months postpartum)" to answer the research question of: "Among women with dysglycemia and a recent history of gestational diabetes mellitus, can acute treatment of semaglutide 1mg lead to regression to normoglycemia?"

ELIGIBILITY:
Inclusion Criteria:

1. Female
2. 18 - 45 years old (inclusive)
3. History of gestational diabetes in most recent pregnancy
4. 6 months - 10 years postpartum
5. BMI ≥ 25 kg/m2
6. Use of long-acting reversible contraception or bilateral tubal ligation
7. Dysglycemia as determined by glycemic response to 75g, 2-hour OGTT: either impaired fasting glucose (IFG), impaired glucose tolerance (IGT), or both (IFG/IGT):

   1. Fasting glucose 100-125mg/dL (inclusive) and/or
   2. 120 minute glucose 140-199mg/dL (inclusive)
8. Willingness to maintain physical activity level throughout study duration
9. Willingness to standardize diet for 3 days prior to OGTT
10. Ability to provide informed consent before any trial-related activities

Exclusion Criteria:

1. Body weight > 350lb
2. Pregnant or the intention of becoming pregnant or not using adequate contraceptive measures.
3. Breastfeeding within 3 months of screening visit 1
4. Post-menopausal
5. Desiring pregnancy within study participation period or two months after participation ends (i.e. 10 months from enrolment)
6. Use of tobacco products within past 6 months
7. Substance or alcohol abuse
8. Presence of significant systemic disease including: diabetes mellitus (type 1 or type 2), cardiac disease (e.g. congestive heart failure), renal impairment (e.g. serum creatinine levels ≥ 1.4 mg/dL or eGFR < 60), hepatic disease (including viral hepatitis, toxic hepatic damage, jaundice of unknown aetiology, or abnormal liver function tests), pancreatitis, uncontrolled thyroid disease (e.g. documented abnormal TSH), adrenal disease (including Cushing's syndrome, congenital adrenal hyperplasia), hyperlipidemia (fasting triglycerides > 399mg%), untreated or poorly controlled hypertension (resting blood pressure >159/94 mmHg)
9. History of or presence of: eating disorder, malignant disease requiring chemotherapy, or debilitating psychiatric disorder such as psychosis or neurological condition that could confound outcome variables
10. History of bariatric surgery
11. Use of medications for glucose regulation: insulin (e.g. Humalog, Novolog, Humulin), pramlintide, metiglinides, metformin, thiazolidinediones, GLP-1 receptor agonists, DPP-4 inhibitors, SGLT2 inhibitors within four weeks of screening visit 1
12. Use of medications for anti-obesity or weight loss within four weeks of screening visit 1
13. Use of medications known to exacerbate glucose dysfunction (such as isotretinoin or corticosteroids) within four weeks of screening visit 1
14. Known or suspected allergy to trial medication, excipients, or related products
15. Contraindications to study medications: patients with a personal or family history of medullary thyroid cancer or in patients with Multiple Endocrine Neoplasia syndrome type 2 (MEN 2)
16. Current or recent past (within 3 months) participation in another experimental drug trial
17. Previous randomization in this trial
18. Receipt of any investigational drug within 6 months prior to this trial

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 102 (Estimated)
Dates: Start 2022-01-13 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Regression to normoglycemia | After 24 weeks of full-dose treatment
  Glucose tolerance to be determined by glycemic response to a 75 gram, two-hour oral glucose tolerance test (OGTT). Regression to normoglycemia is defined by fasting glucose <100mg/dL and 120 minute glucose <140 mg/dL

SECONDARY OUTCOMES:
Change in HbA1c | After 24 weeks of full-dose treatment
  Hemoglobin to be determined
Change in body weight | After 24 weeks of full-dose treatment
  Fasted body weight after intervention minus fasted body weight at enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Sutton, PhD, Principal Investigator — Woman's Hospital, Louisiana
Locations (1):
- Woman's Hospital, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No